CLINICAL TRIAL: NCT03713086
Title: A Non-Randomized, Open Label, Controlled, Dose-Escalation, Phase I Clinical Trial to Evaluate the Safety, Reactogenicity and Immunogenicity of One or Two Administrations of Candidate Rabies mRNA Vaccine CV7202 in Healthy Adult Subjects
Brief Title: A Study to Assess the Safety, Reactogenicity and Immune Response of CureVac's Candidate Rabies mRNA Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV-7202-104; 2017-002856-10 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2022-09

CONDITIONS: Rabies
Keywords: Rabies; Vaccine; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rabipur® (Active Comparator): Participants received 3 doses of Rabipur® intramuscular injection at Days 1, 8 and 29 according to the manufacturer's recommendations.
  Interventions: Biological: Rabipur®
- CV7202 1 mcg (Experimental): Participants received messenger ribonucleic acid (mRNA) CV7202 1 microgram (mcg) intramuscular injection at Day 1, of whom half of the participants received a second dose of CV7202 1 mcg at Day 29.
  Interventions: Biological: Rabies mRNA vaccine CV7202
- CV7202 2 mcg (Experimental): Participants received mRNA CV7202 2 mcg intramuscular injection at Day 1, of whom half of the participants received a second dose of CV7202 2 mcg at Day 29.
  Interventions: Biological: Rabies mRNA vaccine CV7202
- CV7202 5 mcg (Experimental): Participants received mRNA CV7202 5 mcg intramuscular injection at Day 1.
  Interventions: Biological: Rabies mRNA vaccine CV7202

INTERVENTIONS:
Biological: Rabipur® — 3 doses administered IM at Days 1, 8 and 29 in the deltoid region of the arm
  Other Names: Licensed rabies vaccine containing inactivated rabies virus
  Arms: Rabipur®
Biological: Rabies mRNA vaccine CV7202 — CV7202 administered IM at Days 1 and 29 in the deltoid region of the arm
  Arms: CV7202 1 mcg
Biological: Rabies mRNA vaccine CV7202 — CV7202 administered IM at Days 1 and 29 in the deltoid region of the arm
  Arms: CV7202 2 mcg
Biological: Rabies mRNA vaccine CV7202 — CV7202 administered IM at Days 1 and 29 in the deltoid region of the arm
  Arms: CV7202 5 mcg

SUMMARY:
The primary objective of this clinical study is to assess the safety, and reactogenicity of CV7202 mRNA-rabies vaccine in healthy adults. Immunogenicity is also assessed.

ELIGIBILITY:
Inclusion criteria: Subjects must satisfy the following criteria at trial entry:

1. Healthy male and female subjects aged 18 to 40 years inclusive. Healthy Subject is defined as an individual who is in good general health, not having any mental or physical disorder requiring regular or frequent medication.
2. Expected to be compliant with protocol procedures and available for clinical follow-up through the last planned visit.
3. Physical examination and laboratory results without clinically significant findings.
4. Body Mass Index (BMI) ≥18.0 and ≤32.0 kg/m2.
5. Females: At the time of screening, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for women presumed to be of childbearing potential on the day of enrolment. On Day 1 (pre-vaccination): negative urine pregnancy test (hCG), (only required if the screening visit serum pregnancy test was performed more than 3 days before).
6. Females of childbearing potential must use acceptable methods of birth control from 2 weeks before the first administration of the test vaccine until 3 months following the last administration.
7. Males must use reliable forms of contraception (condom) from the moment of the first administration of the test vaccine until 3 months following the last administration and must refrain from sperm donation from the moment of the first administration of the test vaccine until 3 months after the last administration.

Exclusion Criteria Any trial subject who meets any of the following criteria will not qualify for entry into the trial

1. Use of any investigational or non-registered product (drug or vaccine) other than the trial vaccine within 4 weeks preceding the administration of the trial vaccine, or planned use during the trial period.
2. Receipt of any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this trial or planned receipt of any vaccine within 28 days of any trial vaccine administration.
3. Receipt of any licensed or investigational rabies vaccine prior to the administration of the trial vaccine.
4. Planning to travel to regions/countries for which rabies vaccinations are recommended or where high risk of infection exists according to travel recommendations by the German Society of Tropical Medicine and International Health during the trial and up to the end of the trial.
5. Any treatment with immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine or planned use during the trial, with the exception of inhaled and nasal steroids, or topically-applied steroids.
6. Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV) infection and hepatitis C virus (HCV) infection.
7. History of a potential immune mediated disease.
8. Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of any dose of the trial vaccine.
9. Presence or evidence of significant acute or chronic, uncontrolled medical or psychiatric illness.
10. Known allergy to any component of CV7202 such as type I allergy to beta-lactam antibiotics or Rabipur®.
11. Evidence of current alcohol or drug abuse.
12. History of any neurological disorders or seizures including Guillain-Barré syndrome (GBS), with the exception of febrile seizures during childhood.
13. Foreseeable non-compliance with protocol as judged by the investigator.
14. For females: Pregnancy or lactation.
15. History of any life-threatening anaphylactic reactions.
16. Subjects with impaired coagulation or any bleeding disorder in whom an i.m. injection or a blood draw is contraindicated.
17. Known relatives of site research staff working on this trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University Hospital Ghent, Ghent, Belgium
- Department of Infectious Diseases and Tropical Medicine (DITM), Medical Center of the University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Aldrich C, Leroux-Roels I, Huang KB, Bica MA, Loeliger E, Schoenborn-Kellenberger O, Walz L, Leroux-Roels G, von Sonnenburg F, Oostvogels L. Proof-of-concept of a low-dose unmodified mRNA-based rabies vaccine formulated with lipid nanoparticles in human volunteers: A phase 1 trial. Vaccine. 2021 Feb 22;39(8):1310-1318. doi: 10.1016/j.vaccine.2020.12.070. Epub 2021 Jan 22. PMID 33487468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 investigative sites in Germany and Belgium between 12 October 2018 and 23 November 2021.
Pre-assignment Details: A total 90 participants were screened, out of which 53 were enrolled and received the treatment.
Period: Overall Study
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Started | 16 | 16 | 10 | 11
Received Dose at Day 1 | 16 | 16 | 10 | 11
Received Dose at Day 8 | 0 | 0 | 0 | 11
Received Dose at Day 29 | 8 | 8 | 0 | 11
Completed | 16 | 13 | 9 | 10
Not Completed | 0 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data.
Groups:
- CV7202 1 mcg: Participants received mRNA CV7202 1 mcg intramuscular injection at Day 1, of whom half of the participants received a second dose of CV7202 1 mcg at Day 29.
- Total: Total of all reporting groups
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur® | Total
Number analyzed (Participants) | 16 | 16 | 10 | 11 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.62) | 28.3 (5.81) | 26.1 (3.96) | 25.5 (4.23) | 26.9 (5.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 5 | 7 | 33
  Male | 7 | 4 | 5 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 16 | 10 | 11 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 16 | 8 | 10 | 11 | 45
  Germany | 0 | 8 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Local Solicited Adverse Event (AE) Post Dose 1 (Day 1)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Local solicited AEs included injection site pain, redness, swelling, and itching. All AEs were documented in a diary by the participant.
Time Frame: From the first dose of vaccination up to 7 days after vaccination (up to Day 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants | 13 | 15 | 10 | 5

2. Primary Outcome: Number of Participants With Grade 0, 1, 2 and 3 Local Solicited AEs Post Dose 1 (Day 1)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. The intensity of local solicited AEs was graded as:Pain at injection site(Grade 0:absent,Grade 1:Does not interfere with activity, Grade 2:Interferes with activity/repeated use of non-narcotic pain reliever greater than [>] 24 hours,Grade 3:prevent daily activity/repeated use of narcotic pain reliever); Redness(Grade 0:less than or equal to [<=]2.5 centimeters(cm), Grade 1:2.5 to 5cm,Grade 2: 5.1 to 10cm, Grade 3: >10cm);Swelling(Grade 0: <=2.5 cm,Grade 1: 2.5 to 5cm and does not interfere with activity,Grade 2:5.1 to 10cm/interferes with activity,Grade 3:>10cm or prevents daily activity);Itching(Grade 0:absent,Grade 1:Mild,no interference with normal activity,Grade 2:Moderate,some interference with normal activity,Grade 3:Significant, prevents normal activity).
Time Frame: From the first dose of vaccination up to 7 days after vaccination (up to Day 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Grade 0 (No AE/Absent) | 3 | 1 | 0 | 5
  Grade 1 (Mild) | 13 | 13 | 4 | 5
  Grade 2 (Moderate) | 0 | 1 | 5 | 0
  Grade 3 (Severe) | 0 | 1 | 1 | 0
  Not assessed | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants Who Experienced a Systemic Solicited AE and Related Systemic Solicited AE Post Dose 1 (Day 1)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Systemic solicited AEs included fever, nausea/vomiting, diarrhea, headache, fatigue, myalgia, and arthralgia on the day of vaccination and following 7 days after dose 1. All AEs were documented in diary by the participant.
Time Frame: From the first dose of vaccination up to 7 days after vaccination (up to Day 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Participants with Systemic Solicited AE | 11 | 13 | 9 | 8
  Participants with Related Systemic Solicited AE | 8 | 13 | 9 | 5

4. Primary Outcome: Number of Participants With Grade 0, 1, 2, and 3 of Systemic Solicited AEs and Related Systemic Solicited AEs Post Dose 1 (Day 1)
Description: The intensity of Systemic AEs was graded as: Fever(Grade 0: <38 degree Celsius (°C), Grade 1: >=38°C to 38.4°C, Grade 2:>=38.5°C to 38.9°C, Grade 3: >=39°C); Headache(Grade 0: absent, Grade 1: Mild, Grade 2: Moderate, Grade 3: Significant); Fatigue(Grade 0: Absent, Grade 1: Mild, Grade 2: Moderate, Grade 3: Significant); Chills(Grade 0: Absent, Grade 1: Mild, Grade 2: Moderate, Grade 3: Significant); Myalgia(Grade 0: Absent, Grade 1: Mild, Grade 2: Moderate, Grade 3: Significant); Arthralgia(Grade 0: Absent, Grade 1: Mild, Grade 2: Moderate, Grade 3: Significant); Nausea/Vomiting(Grade 0: Absent, Grade 1: Mild, no interference with activity/1-2 episodes/24 hours, Grade 2: Moderate, some interference with activity/>2 episodes/ 24 hours, Grade 3: Severe, prevents daily activity, requires outpatient intravenous [IV] hydration); Diarrhea(Grade 0: Absent, Grade 1: 2-3 stools, Grade 2: 4-5 stools, Grade 3: 6 or more watery stools or requires outpatient IV hydration).
Time Frame: From the first dose of vaccination up to 7 days after vaccination (up to Day 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- CV7202 5 mcg: Participants received mRNA CV7202 5 mcg intramuscular dose at Day 1.
- Rabipur®: Participants received 3 doses of Rabipur® intramuscularly at Days 1, 8 and 29 according to the manufacturer's recommendations.
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Participants with Systemic Solicited AEs: Grade 0 (No AE/Absent) | 5 | 3 | 1 | 2
  Participants with Systemic Solicited AEs: Grade 1 (Mild) | 8 | 4 | 0 | 4
  Participants with Systemic Solicited AEs: Grade 2 (Moderate) | 3 | 6 | 3 | 4
  Participants with Systemic Solicited AEs: Grade 3 (Severe) | 0 | 3 | 6 | 0
  Participants with Systemic Solicited AEs: Not assessed | 0 | 0 | 0 | 1
  Participants with Related Systemic Solicited AEs: Grade 0 (No AE/Absent) | 8 | 3 | 1 | 5
  Participants with Related Systemic Solicited AEs: Grade 1 (Mild) | 5 | 4 | 0 | 2
  Participants with Related Systemic Solicited AEs: Grade 2 (Moderate) | 3 | 6 | 3 | 3
  Participants with Related Systemic Solicited AEs: Grade 3 (Severe) | 0 | 3 | 6 | 0
  Participants with Related Systemic Solicited AEs: Not assessed | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Days of Local Solicited AEs Post Dose 1 (Day 1)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Local solicited AEs included injection site pain, redness, swelling, and itching. All AEs were documented in diary by the participant.
Time Frame: From Day 1 (post-dose 1) to Day 8
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who had an event in the respective category (pain, redness).
Measure: Median (Full Range); unit: Days
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Days
  Pain: number analyzed (Participants) | 13 | 15 | 9 | 5
  Pain | 1 [1 to 4] | 2 [1 to 3] | 3 [1 to 6] | 2 [1 to 4]
  Redness: number analyzed (Participants) | 0 | 0 | 1 | 0
  Redness |  |  | 2 [2 to 2] |

6. Primary Outcome: Number of Days of Local Solicited AEs Post Dose 2
Description: as for outcome 5
Time Frame: CV7202: From Day 29 (post-dose 2) to Day 36; Rabipur: Day 8 (post-dose 2) to Day 15
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | Rabipur®
Number analyzed (Participants) | 8 | 8 | 11
Days
  Pain: number analyzed (Participants) | 5 | 6 | 6
  Pain | 1 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]
  Redness: number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Number of Days of Local Solicited AEs Post Dose 3
Description: as for outcome 5
Time Frame: Day 29 (post-dose 3) to Day 36
Population: as for outcome 5
Measure: Median (Full Range); unit: Days
Arm/Group | Rabipur®
Number analyzed (Participants) | 11
Days
  Pain: number analyzed (Participants) | 5
  Pain | 2 [1 to 2]
  Redness: number analyzed (Participants) | 0

8. Primary Outcome: Number of Days of Systemic Solicited AEs Post Dose 1
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Systemic solicited AEs included fever, nausea/vomiting, chills, diarrhea, headache, fatigue, myalgia, and arthralgia. All AEs were documented in diary by the participant.
Time Frame: From Day 1 (post-dose 1) to Day 8
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who had an event in the respective category (temperature, headache, fatigue, chils, myalgia, arthralgia, nausea/vomiting, diarrhea).
Measure: Median (Full Range); unit: Days
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Days
  Temperature: number analyzed (Participants) | 0 | 3 | 5 | 0
  Temperature |  | 1 [1 to 2] | 1 [1 to 1] |
  Headache: number analyzed (Participants) | 8 | 11 | 7 | 4
  Headache | 1 [1 to 4] | 2 [1 to 5] | 2 [1 to 4] | 1 [1 to 4]
  Fatigue: number analyzed (Participants) | 6 | 9 | 8 | 5
  Fatigue | 2 [1 to 2] | 2 [1 to 3] | 2 [1 to 7] | 1 [1 to 5]
  Chills: number analyzed (Participants) | 0 | 6 | 7 | 0
  Chills |  | 1.5 [1 to 2] | 1 [1 to 2] |
  Myalgia: number analyzed (Participants) | 6 | 7 | 5 | 2
  Myalgia | 2 [1 to 5] | 3 [1 to 3] | 2 [1 to 5] | 1 [1 to 1]
  Athralgia: number analyzed (Participants) | 3 | 3 | 4 | 0
  Athralgia | 1 [1 to 3] | 1 [1 to 2] | 2 [1 to 3] |
  Nausea/Vomiting: number analyzed (Participants) | 1 | 1 | 3 | 1
  Nausea/Vomiting | 1 [1 to 1] | 3 [3 to 3] | 1 [1 to 3] | 1 [1 to 1]
  Diarrhea: number analyzed (Participants) | 1 | 1 | 2 | 0
  Diarrhea | 4 [4 to 4] | 1 [1 to 1] | 2 [1 to 3] |

9. Primary Outcome: Number of Days of Systemic Solicited AEs Post Dose 2
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Systemic solicited AEs included fever, nausea/vomiting, diarrhea, chills, headache, fatigue, myalgia, and arthralgia. All AEs were documented in diary by the participant.
Time Frame: CV7202: From Day 29 (post-dose 2) to Day 36; Rabipur: Day 8 (post-dose 2) to Day 15
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data.
  Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who had an event in the respective category (temperature,headache, fatigue, chills, myalgia, arthralgia, nausea/ vomiting, diarrhea).
Measure: Median (Full Range); unit: Days
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | Rabipur®
Number analyzed (Participants) | 8 | 8 | 11
Days
  Temperature: number analyzed (Participants) | 1 | 2 | 0
  Temperature | 1 [1 to 1] | 1.5 [1 to 2] |
  Headache: number analyzed (Participants) | 4 | 5 | 2
  Headache | 1 [1 to 3] | 2 [1 to 4] | 1.5 [1 to 2]
  Fatigue: number analyzed (Participants) | 4 | 5 | 5
  Fatigue | 2 [1 to 2] | 2 [2 to 3] | 2 [1 to 3]
  Chills: number analyzed (Participants) | 2 | 2 | 0
  Chills | 1.5 [1 to 2] | 1.5 [1 to 2] |
  Myalgia: number analyzed (Participants) | 4 | 5 | 0
  Myalgia | 1.5 [1 to 2] | 1.5 [1 to 2] |
  Arthralgia: number analyzed (Participants) | 3 | 1 | 0
  Arthralgia | 1 [1 to 2] | 2 [2 to 2] |
  Nausea/Vomiting: number analyzed (Participants) | 0 | 1 | 0
  Nausea/Vomiting |  | 2 [2 to 2] |
  Diarrhea: number analyzed (Participants) | 0 | 2 | 0
  Diarrhea |  | 2 [2 to 2] |

10. Primary Outcome: Number of Days of Systemic Solicited AEs Post Dose 3
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Systemic solicited AEs included fever, nausea/vomiting, diarrhea, headache, fatigue, myalgia, and arthralgia. All AEs were documented in diary by the participant.
Time Frame: Day 29 (post-dose 3) to Day 36
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data.
  Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who had an event in the respective category (headache, fatigue, chills).
Measure: Median (Full Range); unit: Days
Arm/Group | Rabipur®
Number analyzed (Participants) | 10
Days
  Headache: number analyzed (Participants) | 3
  Headache | 1 [1 to 1]
  Fatigue: number analyzed (Participants) | 1
  Fatigue | 2 [2 to 2]
  Chills: number analyzed (Participants) | 1
  Chills | 1 [1 to 1]

11. Primary Outcome: Number of Participants Who Experienced Unsolicited and Related Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. An unsolicited AE was defined as any other AE reported by the participant via diary cards or during study visits on the day of vaccination and the 28 subsequent days. The number of participants with unsolicited and related unsolicited AEs were reported.
Time Frame: From the first dose of vaccination up to 28 days after vaccination (up to Day 29)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Participants with Unsolicited AEs | 10 | 14 | 9 | 6
  Participants with Related Unsolicited AEs | 2 | 9 | 7 | 1

12. Primary Outcome: Number of Participants With Grade 1, 2 and 3 Unsolicited and Related Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. An unsolicited AE was defined as any other AE reported by the participant via diary cards or during study visits on the day of vaccination and the 28 subsequent days. The intensity of AEs was graded as: 1) Mild (Grade 1): An event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.; 2) Moderate (Grade 2): An event that caused sufficient discomfort to interfere with normal everyday activities.; 3) Severe (Grade 3): An event that prevented normal everyday activities. Number of participants with Grade 1, 2 and 3 unsolicited and related unsolicited AEs were reported.
Time Frame: From the first dose of vaccination up to 28 days after vaccination (up to Day 29)
Population: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data. Here overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and number analyzed included those participants who were evaluable for the specified categories for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Participants with all unsolicited AEs: number analyzed (Participants) | 10 | 14 | 9 | 6
  Participants with all unsolicited AEs: Grade 1 (Mild) | 3 | 3 | 2 | 2
  Participants with all unsolicited AEs: Grade 2 (Moderate) | 4 | 9 | 1 | 3
  Participants with all unsolicited AEs: Grade 3 (Severe) | 3 | 2 | 6 | 1
  Participants with related unsolicited AEs: number analyzed (Participants) | 2 | 9 | 7 | 1
  Participants with related unsolicited AEs: Grade 1 (Mild) | 1 | 4 | 1 | 0
  Participants with related unsolicited AEs: Grade 2 (Moderate) | 1 | 3 | 1 | 1
  Participants with related unsolicited AEs: Grade 3 (Severe) | 0 | 2 | 5 | 0

13. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs) up to 12 Months
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. SAE was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect.
Time Frame: From the first dose of vaccination up to 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants | 1 | 0 | 0 | 1

14. Primary Outcome: Number of Participants With Any Medically-attended AEs (MAAEs) up to 12 Months
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Vaccine-related MAAEs include any AEs for which the participant received medical attention, defined as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason for which there is evidence to suggest a causal relationship between the study product and the adverse event. Number of participants with any MAAEs were reported.
Time Frame: From the first dose of vaccination up to 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants | 6 | 8 | 3 | 3

15. Primary Outcome: Number of Participants With Any Adverse Events of Special Interest (AESIs) and Related AESI up to 12 Month
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. AEs with a suspected potential immune-mediated disease etiology was considered as AESIs. AESI was assessed by the investigator. Vaccine-related AESIs was included as AESIs for which there was evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: From the first dose of vaccination up to 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
Participants
  Participants with AESIs | 0 | 0 | 0 | 0
  Participants with related AESIs | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Related SAEs From 12 Months Post-vaccination up to 24 Months
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. SAE was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect. Vaccine-related SAEs was included as SAEs for which there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: From 12 months up to 24 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 10
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Related MAAEs From 12 Months up to 24 Months
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. Vaccine-related MAAEs include any AEs for which the participant received medical attention, defined as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason for which there is evidence to suggest a causal relationship between the study product and the adverse event. Number of participants with related MAAEs were reported.
Time Frame: From 12 months up to 24 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 10
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Any Related AESIs From 12 Months up to 24 Months
Description: An AE was defined as any untoward medical occurrence in a clinical study participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. AEs with a suspected potential immune-mediated disease etiology was considered as AESIs. AESI was assessed by the investigator. Vaccine-related AESIs was included as AESIs for which there was evidence to suggest a causal relationship between the study product and the adverse event. Number of participants with any related AESIs were reported.
Time Frame: From 12 months up to 24 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 10
Participants | 0 | 0 | 1 | 0

19. Secondary Outcome: Percentages of Participants With Rabies-specific Serum Virus-neutralizing Antibody Titer (VNTs)
Description: Rabies-specific serum response was defined as VNT ≥ 0.5 international units per milliliter (IU/mL). Rabies-specific serum VNT were measured using the WHO-recommended rapid fluorescent foci inhibition test (RFFIT). Serial dilutions of each serum sample are mixed with a standard dose of rabies virus before tissue culture cells are added. Virus infected cells are detected via a fluorochrome conjugated rabies-specific antibody. If the serum contains antibodies that bind and neutralize the virus, the infectivity of the virus is reduced. The virus neutralization end-point titer is defined as the highest sample dilution at which 50% of the observed microscopic fields contain ≥ 1 infected cell. The percentages of participants with rabies-specific serum VNTs ≥0.5 were taken as positive and were reported.
Time Frame: Baseline (Day 1), Days 15, 43, 365, 547, and 730
Population: Full analysis set (FAS) is a subset of the safety set with participants who had the baseline sample and at least 1 additional blood sample available for VNT analysis. Here overall number of participants analyzed included those participants who were evaluable for this outcome measure and number analyzed included those participants who were evaluable at specified timepoints for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 10
percentage of participants
  Baseline (Day 1) | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]
  Day 15 | 0.0 [0.0 to 20.6] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 30.8] | 100.0 [69.2 to 100.0]
  Day 43: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 43 | 50.0 [24.7 to 75.3] | 62.5 [35.4 to 84.8] | 22.2 [2.8 to 60.0] | 100.0 [69.2 to 100.0]
  Day 365: number analyzed (Participants) | 16 | 14 | 9 | 10
  Day 365 | 12.5 [1.6 to 38.3] | 14.3 [1.8 to 42.8] | 11.1 [0.3 to 48.2] | 100.0 [69.2 to 100.0]
  Day 547: number analyzed (Participants) | 9 | 7 | 6 | 10
  Day 547 | 22.2 [2.8 to 60.0] | 28.6 [3.7 to 71.0] | 16.7 [0.4 to 64.1] | 90.0 [55.5 to 99.7]
  Day 730: number analyzed (Participants) | 9 | 7 | 6 | 10
  Day 730 | 22.2 [2.8 to 60.0] | 42.9 [9.9 to 81.6] | 16.7 [0.4 to 64.1] | 90.0 [55.5 to 99.7]

20. Secondary Outcome: Serum Geometric Mean Titers (GMTs) of Rabies-specific VNTs
Description: Serum geometric mean titer (antilog mean of log-transformed VNTs) was obtained from measuring VNTs using the WHO-recommended rapid fluorescent foci inhibition test. The virus neutralization end-point titer (VNT) is defined as the highest sample dilution at which 50% of the observed microscopic fields contain >=1 infected cell.
Time Frame: Baseline (Day 1), Days 8, 15, 29, 36, 43, 57, 91, 182, 365, 547, and 730
Population: FAS is a subset of the safety set with participants who had the baseline sample and at least 1 additional blood sample available for VNT analysis. Here overall number of participants analyzed included those participants who were evaluable for this outcome measure and number analyzed included those participants who were evaluable at specified timepoints for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: IU/mL
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
Number analyzed (Participants) | 16 | 16 | 10 | 11
IU/mL
  Baseline (Day 1): number analyzed (Participants) | 16 | 16 | 10 | 10
  Baseline (Day 1) | 0.050 (1.0000) | 0.050 (1.0000) | 0.050 (1.0000) | 0.050 (1.0000)
  Day 8: number analyzed (Participants) | 16 | 16 | 10 | 10
  Day 8 | 0.053 (1.2698) | 0.053 (1.2179) | 0.050 (1.0000) | 0.057 (1.3394)
  Day 15: number analyzed (Participants) | 16 | 16 | 10 | 10
  Day 15 | 0.069 (1.8803) | 0.095 (2.6702) | 0.062 (1.5685) | 7.834 (2.7369)
  Day 29: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 29 | 0.092 (1.9864) | 0.189 (3.8604) | 0.144 (2.8064) | 4.478 (3.0074)
  Day 36: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 36 | 0.231 (3.2958) | 0.433 (5.1784) | 0.136 (3.1008) | 8.921 (2.4253)
  Day 43: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 43 | 0.653 (9.3871) | 0.692 (8.3640) | 0.122 (2.9790) | 9.341 (2.2222)
  Day 57: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 57 | 0.540 (8.2728) | 0.502 (7.6846) | 0.125 (2.8786) | 7.849 (1.8818)
  Day 91: number analyzed (Participants) | 16 | 16 | 9 | 10
  Day 91 | 0.445 (5.8568) | 0.275 (6.0428) | 0.105 (2.9133) | 4.888 (1.8755)
  Day 182: number analyzed (Participants) | 15 | 15 | 9 | 10
  Day 182 | 0.176 (4.6498) | 0.163 (3.6199) | 0.074 (2.4421) | 1.089 (1.9244)
  Day 365: number analyzed (Participants) | 16 | 14 | 9 | 10
  Day 365 | 0.095 (2.7511) | 0.097 (2.8842) | 0.072 (2.3457) | 0.816 (2.1405)
  Day 547: number analyzed (Participants) | 9 | 7 | 6 | 10
  Day 547 | 0.132 (2.7428) | 0.149 (3.6318) | 0.077 (2.9198) | 0.879 (1.9594)
  Day 730: number analyzed (Participants) | 9 | 7 | 6 | 10
  Day 730 | 0.128 (3.9213) | 0.246 (4.0963) | 0.073 (2.5600) | 0.831 (2.0624)

ADVERSE EVENTS:
Time Frame: From the first dose of vaccination up to 24 months
Description: Safety analysis set included all participants who had received at least 1 dose of mRNA vaccine CV7202 or Rabipur and those participants who had any post-Day 1 safety data.
Arm/Group | CV7202 1 mcg | CV7202 2 mcg | CV7202 5 mcg | Rabipur®
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 14/16 | 14/16 | 10/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CV7202 1 mcg (N=16) | CV7202 2 mcg (N=16) | CV7202 5 mcg (N=10) | Rabipur® (N=11)
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CV7202 1 mcg (N=16) | CV7202 2 mcg (N=16) | CV7202 5 mcg (N=10) | Rabipur® (N=11)
Nasopharyngitis (Infections and infestations) | 9 | 5 | 7 | 4
Rhinitis (Infections and infestations) | 2 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Strongyloidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 8 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 3 | 0
Chills (General disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1
Influenza like illness (General disorders) | 0 | 3 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0
Injection site warmth (General disorders) | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Oligodipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Allergy to animal (Immune system disorders) | 0 | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Mite allergy (Immune system disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 2
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03713086/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT03713086/SAP_001.pdf